CLINICAL TRIAL: NCT04390893
Title: Comparison of Ultrasound-guided Location of Laryngeal Mask With Air Leakage Test: A Randomized Controlled Trial
Brief Title: Comparison of Ultrasound-guided Location of Laryngeal Mask With Air Leakage Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, ZhiHeng Liu, Head of Anesthesiology Department, Shenzhen Second People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2019-12-07
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Laryngeal Mask
Keywords: ultrasound; air leakage test; bronchofiberscope
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound positioning group (Experimental)
  Interventions: Device: ultrasound
- leak test positioning group (Active Comparator)
  Interventions: Diagnostic Test: air leakage test

INTERVENTIONS:
Device: ultrasound — Anesthesiologist would scan three planes of the neck to position the LMA
  Arms: ultrasound positioning group
Diagnostic Test: air leakage test — Anesthesiologist would use air leakage test to position the LMA
  Arms: leak test positioning group

SUMMARY:
Compare the accuracy of two methods of ultrasound and air leakage test in positioning laryngeal mask. Validate the relationship between ultrasound scores, air leak levels, and bronchoscopic classification in positioning laryngeal mask

ELIGIBILITY:
Inclusion Criteria:

* patients selected for this study must meet all of the following criterion:

  1. Age is between 17 to 65 years old;
  2. ASA (Amecican Society of Anesthesiology ) scores I-II;
  3. Actual weight is between 30 to 100 kilogram;
  4. Patients undergo selective supine operations under general anesthesia (laryngeal mask);
  5. Patients agree to participate in our study and sign Informed Consent Form

Exclusion Criteria:

* Patients cannot participate in this study if they have any of the following conditions:

  1. Airway stenosis, history of airway masses etc, whicn may cause obstruction to ventilation;
  2. Swelling of the neck caused by huge mass in the neck and history of neck surgery etc, which doesn't contribute to ultrasound observation;
  3. Stomach fullness, intestinal obstruction, gastroesophageal reflux disease etc, which may cause reflux aspiration.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound scoring system | during procedure (after laryngeal mask's placement)
  Anesthesiologist who are familiar with ultrasound would scan three planes of neck
Air leakage test grading system | during procedure (after laryngeal mask's placement)
  Anesthesiologist would auscultate the degree of leakage
Fiberoptic scoring system | procedure (after ultrasound examination or leakage test)
  Anesthesiologist would confirm the position of LMA by fiberscope

SECONDARY OUTCOMES:
Complications related to LMA (laryngeal mask airway ) | 24 hours after surgery
  such as reflection of tussis, sore throat, hoarseness, bleeding and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Song K, Yi J, Liu W, Huang S, Huang Y. Confirmation of laryngeal mask airway placement by ultrasound examination: a pilot study. J Clin Anesth. 2016 Nov;34:638-46. doi: 10.1016/j.jclinane.2016.06.019. Epub 2016 Aug 3. PMID 27687463
- [Result] Perez-Herrero MA, de la Varga O, Flores M, Sanchez-Ruano J, Otero M, Buisan F. Descriptive study of ultrasound images of the upper airway obtained after insertion of laryngeal mask. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Oct;65(8):434-440. doi: 10.1016/j.redar.2018.05.004. Epub 2018 Jun 30. English, Spanish. PMID 29970248
- [Result] Osman A, Sum KM. Role of upper airway ultrasound in airway management. J Intensive Care. 2016 Aug 15;4:52. doi: 10.1186/s40560-016-0174-z. eCollection 2016. PMID 27529028
- [Result] Zhou ZF, Xia CZ, Wu M, Yu LN, Yan GZ, Ren QS, Hu CX, Yan M. Comparison of three methods for the confirmation of laryngeal mask airway placement in female patients undergoing gynecologic surgery. Ultrasound Med Biol. 2015 May;41(5):1212-20. doi: 10.1016/j.ultrasmedbio.2014.12.002. Epub 2015 Mar 5. PMID 25748523
- [Result] Kim J, Kim JY, Kim WO, Kil HK. An ultrasound evaluation of laryngeal mask airway position in pediatric patients: an observational study. Anesth Analg. 2015 Feb;120(2):427-32. doi: 10.1213/ANE.0000000000000551. PMID 25545750
- [Result] Ghai B, Ram J, Makkar JK, Wig J. Fiber-optic assessment of LMA position in children: a randomized crossover comparison of two techniques. Paediatr Anaesth. 2011 Nov;21(11):1142-7. doi: 10.1111/j.1460-9592.2011.03632.x. Epub 2011 Jun 21. PMID 21689206